CLINICAL TRIAL: NCT05616923
Title: Topical Mitogenic-Activated Protein Kinase (MAPK) Inhibition in Rosacea
Acronym: TOMIR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albany Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 137506
Record Dates: First submitted 2022-11-09; First posted 2022-11-15 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Rosacea, Erythematotelangiectatic
MeSH Terms: conditions — Rosacea | interventions — trametinib; p38 MAPK inhibitor SB203582

STUDY DESIGN:
Intervention Model Description: Each patient will receive two creams labeled "right cheek" or "left cheek", one containing the active ingredient and the other serving as vehicle control. The labels of each bottle were randomized and the contents of each remains blinded to both the subject and the investigator.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation of drug to cheek side for each bottle set is known only to an investigator not involved in patient assessment and will be unmasked only at the end of the trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trametinib (Experimental): Cheek describing the active compound (topical cream containing 0.1 mg/g trametinib)
  Interventions: Drug: Trametinib
- Vehicle (Placebo Comparator): Cheek receiving cream without active compound (topical cream lacking active ingredient)
  Interventions: Drug: Trametinib

INTERVENTIONS:
Drug: Trametinib — Topical cream containing 0.1 mg/g trametinib
  Other Names: MAPK inhibitor

SUMMARY:
This is a prospective, vehicle controlled, double blinded study to evaluate the safety and potential efficacy of a topical formulation of a MEK inhibitor in patients with erythematotelangiectatic rosacea

DETAILED DESCRIPTION:
The duration of the study will be 22 days. Subjects will use a cream with a mitogen-activated extracellular signal-regulated kinase (MEK) inhibitor on one cheek, and a cream lacking the inhibitor (vehicle control) on the other. Patients will receive a randomized set of creams for the right and left cheek, one containing the active ingredient. Subjects will be evaluated on days 1, 8, 15 and 22. Skin appearance will be scored in each visit. A blood sample will be obtained to determine the levels of systemic drug absorption.

ELIGIBILITY:
Inclusion Criteria:

* Erythematotelangiectatic rosacea diagnosed by a clinician in the centrofacial and/or ocular regions.

Exclusion Criteria:

* Other concurrent diseases for which treatment is being received that would preclude the use of trametinib (i.e., pleural effusion, active infection, intracranial bleeding)
* History of skin allergic reactions or documented allergic reaction to trametinib
* Pregnancy or lactation.
* Heart failure or other heart disease
* Active use of medications with known documented interactions with trametinib (Chloroquine, Ritonavir, Loperamide, Penicillamine)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in dermatologic score | 22 days
  Weekly assessment of skin irritation, using the Organization for Economic Cooperation and Development test for dermal irritation and corrosion. This test measures cutaneous erythema and edema separately on scales that range from 0 (absence of erythema or edema) to 4 (severe), with higher scores representing worse outcomes.

SECONDARY OUTCOMES:
Systemic drug absorption | 22 days
  Blood levels of trametinib will be assessed by high-performance liquid chromatography

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Busingye, MD, Principal Investigator — Stratton VA Medical Center
Locations (1):
- Samuel S. Stratton VA Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No